CLINICAL TRIAL: NCT04917783
Title: Health Literacy: A Randomized Controlled Trial to Investigate a Novel Feedback Tool for Neurocognitive Screening in Pediatric Sickle Cell Disease
Brief Title: Health Literacy - Neurocognitive Screening in Pediatric SCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Jeffrey Karst, Assistant Professor of Pediatrics, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1345169
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Sickle Cell Disease
Keywords: Health Literacy; Neuropsychology; Hematology; academic achievement
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Investigator
Masking Description: This study will use a single-blinded (qualitative coder), randomized controlled trial to evaluate the efficacy of the passport card in improving caregiver understanding and follow through with testing recommendations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Other): Caregivers in the standard of care-arm will receive immediate verbal feedback by a psychologist on their neurocognitive testing results, recommendations, and guidance for implementing recommendations (e.g., sending a 504 Plan request to the school). This report will contain information regarding background, test results, a summary and impressions, and bullet-pointed recommendations.
  Interventions: Behavioral: No Passport card
- Health Literacy (Experimental): Participants randomized to the experimental health-literacy group will be provided with a color-coded "passport" (a two-sided wallet-sized card) highlighting key findings and recommendations of their neurocognitive testing results along with the full written report. The domains listed as either satisfactory or needing help listed on the passport card will directly correspond to those listed on the full report.
  Interventions: Behavioral: Passport Card

INTERVENTIONS:
Behavioral: Passport Card — After receiving neurocognitive testing, caregivers in the health-literacy group will be provided with a color-coded "passport" (a two-sided wallet-sized card) highlighting key findings and recommendations along with their written report. Then, approximately 7 - 14 weeks after testing, caregivers will complete a brief questionnaire in person during their follow-up clinic visit or via phone if necessary. The person completing the parent/caregiver/guardian report must have been present for the evaluation and feedback session and must be the parent/caregiver/guardian who received the feedback passport card and evaluation report.
  Arms: Health Literacy
Behavioral: No Passport card — After receiving neurocognitive testing and verbal feedback from the psychologist, approximately 7 - 14 weeks after testing, caregivers will complete a brief questionnaire in person during their follow-up clinic visit or via phone if necessary. The person completing the parent/caregiver/guardian report must have been present for the evaluation and feedback session and must be the parent/caregiver/guardian who received the feedback and evaluation report, but not the passport card.
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to determine feasibility and potential benefits of providing a passport card with a summary of neurocognitive feedback results to families of patients with sickle cell disease. Given recent literature suggesting the need to be conscious of health literacy in populations with low socioeconomic status, this project is intended to provide a more health-literate appropriate format of neurocognitive evaluation feedback in the context of a routine screening program offered as a standard of care in the CHW pediatric sickle cell disease clinic. The specific aims is (1) to evaluate differences in caregiver understanding of neurocognitive report findings when provided with a health-literate passport card compared to control group and (2) to evaluate differences in follow-through on neurocognitive report recommendations when provided with a health-literate passport card compared to control group.

DETAILED DESCRIPTION:
Pediatric sickle cell disease (SCD) is a blood disorder affecting approximately 70,000 to 100,000 individuals in the United States. Approximately 80% of individuals affected by SCD are African American, with approximately one out of every 346 individuals in this racial group diagnosed. Sickle cell disease is associated with broad neurocognitive impairment. Compared to their healthy peers, children with SCD demonstrate deficits in intellectual functioning, verbal abilities, visual-motor, and visual-spatial skills, short-term memory, executive functioning, attention and focus, and processing speed.

Neurocognitive deficits can result from primary disease-related factors including chronic anemia, hypoxemia, or cerebrovascular ischemia; as well as secondary factors such as missed school and a higher prevalence of socio-economic disadvantages in African American children. While direct neurological impact appears to be associated with neurocognitive performance, it was found that even children with no MRI abnormality evidence lower intellectual functioning skills than healthy controls, suggesting that "biological, socioeconomic, and environmental" factors are all implicated in neurocognitive impairment.

Because of these deficits, children with SCD are more likely to be retained in school relative to other African American students at the local and national levels. In addition, poorer cognitive and academic performance is associated with a decrease in patient-reported quality of life and general psychosocial functioning. In turn, greater levels of stress and negative mood are correlated with higher levels of reported pain, greater health care utilization, and reduced physical activity. It appears that sickle cell disease not only contributes to poorer neurocognitive and social-emotional well-being, but that declines in these domains can further exacerbate sickle cell disease symptoms.

Because of the deficits in neurocognitive functioning of children with SCD, routine screening is recommended to assess for cognitive deficits and provide appropriate recommendations. Unfortunately, prior research in SCD suggests limited follow-up on referrals and recommendations. For example, it was found that 25% of children with SCD evaluated by a neuropsychologist met the criteria for ADHD, but only 21% of the children subsequently diagnosed with ADHD were prescribed medication. In addition, it was found that children with SCD were not universally receiving appropriate school accommodations and interventions based on their cognitive deficits, despite the recommendation that school-based services be implemented immediately for children with SCD.

The disconnect between the cognitive, emotional/behavioral, and academic deficits are typically seen in children with SCD and the actual support received may be due in part to low health literacy and the provision of complex reports following testing. Health literacy has been found to be low in adolescents and adults with sickle cell disease. Another study found that caregivers of children with SCD had a low level of baseline disease-related knowledge but that this knowledge did improve with in-person education; however, this knowledge appeared to decline over time. Unfortunately, materials developed to improve knowledge often do not fit criteria for broad population health literacy. One study found that patient education materials developed for patients with sickle cell disease and their families ranged from an 8th to 12th grade reading level, with limited potential to translate written recommendations into concrete actions.

Broadly, research suggests the need for a change within the historical format of neurocognitive evaluation reports. It is noted as a need to make written reports provided to families more efficient, readable, and effective. Providing appropriate feedback to families appears essential, as it can improve health-related quality of life, coping, and understanding. An informal calculation of the current reports provided to families in our clinic's neurocognitive screening program suggested that reports averaged a reading level grade of 12.3 and approximately 17,500 words, standing in stark contrast to health literacy recommendations. Addressing the poor health literacy of neurocognitive feedback evaluations has two primary problems. First, these reports often have multiple intended audiences beyond caregivers, including teachers, school psychologists, physicians, and other professionals working with the child. These individuals may benefit from more detailed and technical information. In addition, some of the wording used in neurocognitive reports is standardized and can lose meaning or be technically incorrect if simplified. Thus, it appears essential to evaluate whether the addition of a health-literate passport card will help address disparities in understanding of results and patient/family follow-through after receiving a neurocognitive evaluation.

This study is innovative in being the first to our knowledge to investigate the use of a tangible tool, namely a "passport" style printed card, to address health literacy concerns by conveying the most important findings and recommended follow-up after completion of a neurocognitive evaluation. In other contexts, healthcare passport cards have demonstrated the ability to improve communication among families and other providers, make information and recommendations portable, and enhance continuity of care. However, the use of passport cards has not been evaluated as a potential solution to the problem plaguing neuropsychological evaluations, namely the provision of overly lengthy and complex reports following testing.

ELIGIBILITY:
Inclusion Criteria:

* Participants will include English-speaking patients between the ages of 6 and 17 with pediatric sickle cell disease and their caregivers (46 patient-caregiver dyads).

Exclusion Criteria:

* Patients will be excluded from participation if they have a history of significant neurological injury or impairment negating the benefit of a neurocognitive screening

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Caregiver Understanding | 7-14 weeks post evaluation
  Evaluate differences in caregiver understanding of neurocognitive report findings when provided with a health-literate passport card compared to the control group through the semi-structured interview.
Caregiver Follow-through | 7-14 weeks post evaluation
  Evaluate differences in follow-through on neurocognitive report recommendations when provided with a health-literate passport card compared to the control group through the semi-structured interview.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Karst, PhD, Principal Investigator — Medical College of Wisconsin
Locations (2):
- United States (2):
  - Children's Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
As of right now we are not going to share study documents or data.

REFERENCES:
- [Background] Acquazzino MA, Miller M, Myrvik M, Newby R, Scott JP. Attention Deficit Hyperactivity Disorder in Children With Sickle Cell Disease Referred for an Evaluation. J Pediatr Hematol Oncol. 2017 Jul;39(5):350-354. doi: 10.1097/MPH.0000000000000847. PMID 28538513
- [Background] Anie KA. Psychological complications in sickle cell disease. Br J Haematol. 2005 Jun;129(6):723-9. doi: 10.1111/j.1365-2141.2005.05500.x. PMID 15952997
- [Background] Baum KT, von Thomsen C, Elam M, Murphy C, Gerstle M, Austin CA, Beebe DW. Communication is key: the utility of a revised neuropsychological report format. Clin Neuropsychol. 2018 Apr;32(3):345-367. doi: 10.1080/13854046.2017.1413208. Epub 2017 Dec 15. PMID 29243544
- [Background] Berkelhammer LD, Williamson AL, Sanford SD, Dirksen CL, Sharp WG, Margulies AS, Prengler RA. Neurocognitive sequelae of pediatric sickle cell disease: a review of the literature. Child Neuropsychol. 2007 Mar;13(2):120-31. doi: 10.1080/09297040600800956. PMID 17364569
- [Background] Brandow AM, Zappia KJ, Stucky CL. Sickle cell disease: a natural model of acute and chronic pain. Pain. 2017 Apr;158 Suppl 1(Suppl 1):S79-S84. doi: 10.1097/j.pain.0000000000000824. No abstract available. PMID 28221286
- [Background] Caldwell EP, Carter P, Becker H, Mackert M. The Use of the Newest Vital Sign Health Literacy Instrument in Adolescents With Sickle Cell Disease. J Pediatr Oncol Nurs. 2018 Sep/Oct;35(5):361-367. doi: 10.1177/1043454218767875. Epub 2018 Apr 16. PMID 29658377
- [Background] Creary S, Adan I, Stanek J, O'Brien SH, Chisolm DJ, Jeffries T, Zajo K, Varga E. Sickle cell trait knowledge and health literacy in caregivers who receive in-person sickle cell trait education. Mol Genet Genomic Med. 2017 Nov;5(6):692-699. doi: 10.1002/mgg3.327. Epub 2017 Aug 23. PMID 29178654
- [Background] Daly, B. P., Kral, M. C., & Brown, R. T. (2008). Cognitive and academic problems associated with childhood cancers and sickle cell disease. School Psychology Quarterly, 23(2), 230-242. https://doi.org/10.1037/1045-3830.23.2.230
- [Background] Davis DW, Jones VF, Logsdon MC, Ryan L, Wilkerson-McMahon M. Health promotion in pediatric primary care: importance of health literacy and communication practices. Clin Pediatr (Phila). 2013 Dec;52(12):1127-34. doi: 10.1177/0009922813506607. Epub 2013 Oct 21. PMID 24146229
- [Background] Gil KM, Carson JW, Porter LS, Ready J, Valrie C, Redding-Lallinger R, Daeschner C. Daily stress and mood and their association with pain, health-care use, and school activity in adolescents with sickle cell disease. J Pediatr Psychol. 2003 Jul-Aug;28(5):363-73. doi: 10.1093/jpepsy/jsg026. PMID 12808013
- [Background] Hardy SJ, Bills SE, Wise SM, Hardy KK. Cognitive Abilities Moderate the Effect of Disease Severity on Health-Related Quality of Life in Pediatric Sickle Cell Disease. J Pediatr Psychol. 2018 Sep 1;43(8):882-894. doi: 10.1093/jpepsy/jsy019. PMID 29659914
- [Background] Haywood C Jr, Lanzkron S, Ratanawongsa N, Bediako SM, Lattimer L, Powe NR, Beach MC. The association of provider communication with trust among adults with sickle cell disease. J Gen Intern Med. 2010 Jun;25(6):543-8. doi: 10.1007/s11606-009-1247-7. Epub 2010 Mar 3. PMID 20195785
- [Background] Kawadler JM, Clayden JD, Clark CA, Kirkham FJ. Intelligence quotient in paediatric sickle cell disease: a systematic review and meta-analysis. Dev Med Child Neurol. 2016 Jul;58(7):672-9. doi: 10.1111/dmcn.13113. Epub 2016 Mar 31. PMID 27038278
- [Background] Kral MC, Brown RT, Hynd GW. Neuropsychological aspects of pediatric sickle cell disease. Neuropsychol Rev. 2001 Dec;11(4):179-96. doi: 10.1023/a:1012901124088. PMID 11883668
- [Background] McCleary-Jones V. Health literacy and its association with diabetes knowledge, self-efficacy and disease self-management among African Americans with diabetes mellitus. ABNF J. 2011 Spring;22(2):25-32. PMID 21675666
- [Background] McClure E, Ng J, Vitzthum K, Rudd R. A Mismatch Between Patient Education Materials About Sickle Cell Disease and the Literacy Level of Their Intended Audience. Prev Chronic Dis. 2016 May 12;13:E64. doi: 10.5888/pcd13.150478. PMID 27172259
- [Background] Morrison AK, Myrvik MP, Brousseau DC, Drendel AL, Scott JP, Visotcky A, Panepinto JA. Parents' pain medication underdosing is associated with more emergency department visits in sickle cell disease. Pediatr Blood Cancer. 2018 Apr;65(4):10.1002/pbc.26906. doi: 10.1002/pbc.26906. Epub 2017 Dec 12. PMID 29230919
- [Background] Nobile C, Drotar D. Research on the quality of parent-provider communication in pediatric care: implications and recommendations. J Dev Behav Pediatr. 2003 Aug;24(4):279-90. doi: 10.1097/00004703-200308000-00010. PMID 12915801
- [Background] Noll RB, Stith L, Gartstein MA, Ris MD, Grueneich R, Vannatta K, Kalinyak K. Neuropsychological functioning of youths with sickle cell disease: comparison with non-chronically ill peers. J Pediatr Psychol. 2001 Mar;26(2):69-78. doi: 10.1093/jpepsy/26.2.69. PMID 11181883
- [Background] Ohene-Frempong K, Weiner SJ, Sleeper LA, Miller ST, Embury S, Moohr JW, Wethers DL, Pegelow CH, Gill FM. Cerebrovascular accidents in sickle cell disease: rates and risk factors. Blood. 1998 Jan 1;91(1):288-94. PMID 9414296
- [Background] Perry EL, Carter PA, Becker HA, Garcia AA, Mackert M, Johnson KE. Health Literacy in Adolescents With Sickle Cell Disease. J Pediatr Nurs. 2017 Sep-Oct;36:191-196. doi: 10.1016/j.pedn.2017.05.012. Epub 2017 Jul 7. PMID 28888502
- [Background] Rosado DL, Buehler S, Botbol-Berman E, Feigon M, Leon A, Luu H, Carrion C, Gonzalez M, Rao J, Greif T, Seidenberg M, Pliskin NH. Neuropsychological feedback services improve quality of life and social adjustment. Clin Neuropsychol. 2018 Apr;32(3):422-435. doi: 10.1080/13854046.2017.1400105. Epub 2017 Nov 8. PMID 29115189
- [Background] Routhieaux J, Sarcone S, Stegenga K. Neurocognitive sequelae of sickle cell disease: current issues and future directions. J Pediatr Oncol Nurs. 2005 May-Jun;22(3):160-7. doi: 10.1177/1043454205275408. PMID 15855477
- [Background] Schatz J, Brown RT, Pascual JM, Hsu L, DeBaun MR. Poor school and cognitive functioning with silent cerebral infarcts and sickle cell disease. Neurology. 2001 Apr 24;56(8):1109-11. doi: 10.1212/wnl.56.8.1109. PMID 11320190
- [Background] Steen RG, Fineberg-Buchner C, Hankins G, Weiss L, Prifitera A, Mulhern RK. Cognitive deficits in children with sickle cell disease. J Child Neurol. 2005 Feb;20(2):102-7. doi: 10.1177/08830738050200020301. PMID 15794173
- [Background] Weekes CV. African Americans and health literacy: a systematic review. ABNF J. 2012 Fall;23(4):76-80. PMID 23311265
- [Background] Williams AM, Zent CS, Janelsins MC. What is known and unknown about chemotherapy-related cognitive impairment in patients with haematological malignancies and areas of needed research. Br J Haematol. 2016 Sep;174(6):835-46. doi: 10.1111/bjh.14211. Epub 2016 Jul 8. PMID 27391367
- [Background] Wills KE, Nelson SC, Hennessy J, Nwaneri MO, Miskowiec J, McDonough E, Moquist K. Transition planning for youth with sickle cell disease: embedding neuropsychological assessment into comprehensive care. Pediatrics. 2010 Dec;126 Suppl 3:S151-9. doi: 10.1542/peds.2010-1466J. PMID 21123479
- [Background] Yawn BP, Buchanan GR, Afenyi-Annan AN, Ballas SK, Hassell KL, James AH, Jordan L, Lanzkron SM, Lottenberg R, Savage WJ, Tanabe PJ, Ware RE, Murad MH, Goldsmith JC, Ortiz E, Fulwood R, Horton A, John-Sowah J. Management of sickle cell disease: summary of the 2014 evidence-based report by expert panel members. JAMA. 2014 Sep 10;312(10):1033-48. doi: 10.1001/jama.2014.10517. PMID 25203083
- [Background] Schatz J, Finke R, Roberts CW. Interactions of biomedical and environmental risk factors for cognitive development: a preliminary study of sickle cell disease. J Dev Behav Pediatr. 2004 Oct;25(5):303-10. doi: 10.1097/00004703-200410000-00001. PMID 15502546
- [Background] Daly B, Kral MC, Tarazi RA. The role of neuropsychological evaluation in pediatric sickle cell disease. Clin Neuropsychol. 2011 Aug;25(6):903-25. doi: 10.1080/13854046.2011.560190. PMID 21563016